CLINICAL TRIAL: NCT02756949
Title: Do Smartphones Increase Linkage to and Retention in Care in Newly Diagnosed HIV-positive Patients in Johannesburg, South Africa: A Multisite Randomised Controlled Trial
Brief Title: Smart Linkage-to-HIV Care Via a Smartphone App
Acronym: SmartLtC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Bank (Other)
Collaborators: Wits Reproductive Health and HIV Institute (Other); National Health Laboratory Service South Africa (Unknown); Department for International Development, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7173708
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Results first posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-04

CONDITIONS: HIV Infections; Viral Load; Patient Compliance; Antiretroviral Therapy; Cell Phone
Keywords: HIV; Viral load; CD4 count; mHealth; Smartphone; Linkage to care; Retention in care; Antiretroviral treatment; Randomized controlled trial; Johannesburg; Mobile app; Treatment adherence
MeSH Terms: conditions — HIV Infections; Patient Compliance; Treatment Adherence and Compliance | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smartphone-enabled app for linkage to care (Experimental): Participants in this arm are randomised to receive the smartphone application which provides direct access to HIV-related laboratory test results.
  Interventions: Other: Smartphone application; Device: Smartphone
- Standard of care (No Intervention): Participants in this arm are randomised to receive standard of care services.

INTERVENTIONS:
Other: Smartphone application — Laboratory result data will be presented in the app with simple explanations on every screen. English and Zulu languages will be offered in the same app and written at a grade 4 reading level (as per WHO guidelines on literacy). Laboratory results will be supplemented with informative and relevant information explaining the result that has been shown and the recommended action for the patient to take. Patients will also be able to view additional HIV-related information and a Frequently Asked Questions (FAQ) through the app.
  Other Names: App; Customised smartphone app
  Arms: Smartphone-enabled app for linkage to care
Device: Smartphone
  Arms: Smartphone-enabled app for linkage to care

SUMMARY:
This randomized controlled trial evaluates the provision of individual patient laboratory results to newly diagnosed HIV positive smartphone users through a secure application (app) as a method to get them linked to and retained in care, and engage with educational materials purposefully developed to explain their results. Message prompts will also be used to alert patients that their results are ready and provide information on how to link to care, and assistance to re-link to care if they fall out of the health system for any reason. Prompts will be sent to patients to remind health care workers if they are due for repeat laboratory monitoring. The primary endpoint is linkage to care (a HIV-related laboratory test) at 6 months. The control group received standard of care.

DETAILED DESCRIPTION:
This evaluation of a newly designed smartphone application (app) for linkage to care, HIV treatment adherence and retention in care, is taking place at five Johannesburg health facilities. Intervention allocation is random with individuals either receiving the smartphone app or standard of care. The trial is motivated by evidence from elsewhere that sending lab results via app acceptable, and loss of patients in need of HIV care can be reduced with mobile Health interventions. There is a growing number of smartphones in South Africa (at the time of baseline assessment, about 40% of the surveyed population had an Android smartphone with data, and the majority of new phones are smartphones). The trial's objectives are: a) Test whether routine linkage to HIV care at public sector services is improved by providing HIV positive clients with a smartphone-enabled app when compared to standard of care; b) Determine HIV treatment initiation rates between intervention and control arm; c) Test the feasibility and acceptability of receiving lab results via app; d) Assess secondary effects from improved participant information, including return rates after falling out of care, participant satisfaction, and rates of repeat blood tests; e) Determine knowledge levels on HIV care; and f) Assess the effect in priority groups for better linkage to care (male HIV cases and HIV positive youth). If data allow, a cost-benefit analysis will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed HIV positive clients presenting at selected public health facilities, irrespective of CD4 count
* Access to an Android smartphone with data
* Willing to pay the (very small) cost to access their laboratory result
* Age - 18 years and older
* Proof of ID/passport/refugee number (for identification/security, and to confirm the single patient identifier)
* Can read English or Zulu
* Ability and willingness to sign informed consent

Exclusion Criteria:

* Clients presenting for antenatal care services, as these women will be enrolled in the national MomConnect program
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Venter, Prof, Study Director — Wits Reproductive Health and HIV Institute
Locations (1):
- Wits Reproductive Health and HIV Institute, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Venter WDF, Fischer A, Lalla-Edward ST, Coleman J, Lau Chan V, Shubber Z, Phatsoane M, Gorgens M, Stewart-Isherwood L, Carmona S, Fraser-Hurt N. Improving Linkage to and Retention in Care in Newly Diagnosed HIV-Positive Patients Using Smartphones in South Africa: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Apr 2;7(4):e12652. doi: 10.2196/12652. PMID 30938681
- [Result] Venter W, Coleman J, Chan VL, Shubber Z, Phatsoane M, Gorgens M, Stewart-Isherwood L, Carmona S, Fraser-Hurt N. Improving Linkage to HIV Care Through Mobile Phone Apps: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Jul 17;6(7):e155. doi: 10.2196/mhealth.8376. PMID 30021706
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- See also: Smart Linkage to Care : Evaluation Report — http://hdl.handle.net/10986/30862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 5 public HIV testing sites (1 community health center, 3 clinics, and 1 tertiary hospital) in inner city Johannesburg, South Africa. Recruitment happened from October 2015 to June 2016. HIV positive individuals were pre-screened for trial suitability and recruited if eligible upon screening.
Pre-assignment Details: Of the 4537 individuals approached about the study, 90 declined to participate and 4094 were found ineligible during pre-screening and screening, leaving 353 for randomization. 8 standard of care arm participants were later removed from analysis due to erroneous sending of SMS reminders for their 6-month clinic appointment leaving 345 for analysis.
Groups:
- Smartphone-enabled App for Linkage to Care: Participants in this arm are randomised to receive the smartphone application which provides direct access to HIV-related laboratory test results.
  Smartphone application: Laboratory result data will be presented in the app with simple explanations on every screen. English and Zulu languages will be offered in the same app and written at a grade 4 reading level (as per WHO guidelines on literacy). Laboratory results will be supplemented with informative and relevant information explaining the result that has been shown and the recommended action for the patient to take. Patients will also be able to view additional HIV-related information and a Frequently Asked Questions (FAQ) through the app.
  Smartphone
Period: Overall Study
Arm/Group | Smartphone-enabled App for Linkage to Care | Standard of Care
Started | 181 | 172
Completed | 181 | 164
Not Completed | 0 | 8

BASELINE CHARACTERISTICS:
Population: 35% of the participants were male and 44% were aged 18-29 years. 48% of participants were employed full time and 96% had at least attended secondary school. 57% were South Africa born and 36% Zimbabwean. The 2 trial arms were well balanced for these participants' characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Smartphone-enabled App for Linkage to Care | Standard of Care | Total
Number analyzed (Participants) | 181 | 164 | 345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 181 | 164 | 345
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 103 | 224
  Male | 60 | 61 | 121
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Africa | 181 | 164 | 345
Country of birth [Count of Participants; unit: Participants] — Population: Eight participants in the control arm were removed from analysis due to erroneous sending of SMS message to them leading to a contamination issue.
  Participants | 181 | 164 | 345
Education level [Count of Participants; unit: Participants] — Primary only, Some secondary, Completed secondary, attended/completed tertiary Population: Eight control arm participants excluded due to contamination of intervention
  Participants
    Primary only | 8 | 6 | 14
    Some secondary school | 51 | 44 | 95
    Completed secondary school | 98 | 85 | 183
    Attended/completed tertiary | 24 | 29 | 53
Employment status [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Eight control arm participants excluded due to contamination of intervention
  Participants
    Full time | 82 | 79 | 161
    Part time | 37 | 22 | 59
    Unemployed | 49 | 40 | 89
    Self-employed | 10 | 16 | 26
    Student | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Linkage to HIV Care (Indicated by a HIV-related Laboratory Blood Test Within 8 Months)
Description: To test whether linkage to HIV care is improved by providing new HIV clients with access to a smartphone-enabled application (app) when compared to standard of care around 6 months post-diagnosis.
Time Frame: Recruitment +8 months
Population: Eight standard of care participants removed from analysis due to contamination of the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Smartphone-enabled App for Linkage to Care | Standard of Care
Number analyzed (Participants) | 181 | 164
Participants
  Linked to HIV care | 88 | 74
  Not linked | 93 | 90

2. Secondary Outcome: Linkage to HIV Care Among Young People (Indicated by a HIV-related Laboratory Blood Test Within 8 Months)
Description: To test whether among individuals aged 18-30 years linkage to HIV care is improved by providing new HIV clients with access to a smartphone-enabled application (app) when compared to standard of care around 6 months post-diagnosis.
Time Frame: Recruitment +8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Smartphone-enabled App for Linkage to Care | Standard of Care
Number analyzed (Participants) | 83 | 69
Participants
  Linked to HIV care | 44 | 22
  Not linked | 39 | 47

ADVERSE EVENTS:
Time Frame: 12 months
Description: Since this was an intervention testing a smartphone app and not a medical intervention as such, adverse event monitoring was not part of the trial. However, we would have recorded death of a study participant in case a death had occurred.
Arm/Group | Smartphone-enabled App for Linkage to Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/164
Serious Adverse Events (participants affected / at risk) | 0/181 | 0/164
Other Adverse Events (participants affected / at risk) | 0/181 | 0/164

LIMITATIONS AND CAVEATS:
ART initiation, participant satisfaction, knowledge scores) could not be evaluated. Analytics on app use could not be conducted. Generalization of findings is limited due to smart phone requirement for trial participation (selection bias).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT02756949/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2015-05-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT02756949/Prot_ICF_001.pdf